CLINICAL TRIAL: NCT01893034
Title: A Randomised Controlled Trial of Surgical Versus Non-surgical Treatment of Femoroacetabular Impingement
Brief Title: Trial for Femoroacetabular Impingement Treatment
Acronym: FAIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAIT
Record Dates: First submitted 2013-06-14; First posted 2013-07-08 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Femoroacetabular Impingement
Keywords: Femoroacetabular Impingement; Arthroscopy; Physiotherapy; Randomised Controlled Trial
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Physical Therapy Modalities

ARMS (2):
- Conservative treatment (Active Comparator): Physiotherapy and activity modification
  Interventions: Other: Physiotherapy and activity modification
- Surgical treatment (Active Comparator): Arthroscopic treatment of femoroacetabular impingement
  Interventions: Procedure: Arthroscopic treatment of femoroacetabular impingement

INTERVENTIONS:
Procedure: Arthroscopic treatment of femoroacetabular impingement
  Arms: Surgical treatment
Other: Physiotherapy and activity modification
  Arms: Conservative treatment

SUMMARY:
Femoroacetabular Impingement (FAI) describes a condition of the hip where additional bone results in the abutment of the femoral neck against the rim of the acetabulum. This gives rise to localised cartilage damage and pain, but also increases the risk of developing osteoarthritis. The purpose of this study is to compare the effectiveness of arthroscopic surgery versus physiotherapy and activity modification for the treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients
* Age 18-60 years
* Clinical and radiological evidence of FAI
* Competent to consent

Exclusion Criteria:

* Prior hip surgery
* Established osteoarthritis (Kellgren-Lawrence >/= 2)
* Hip dysplasia (Centre-Edge angle < 20 degrees on radiograph)
* Completion of physiotherapy programme targeting FAI within past year
* Co-morbidities that mean surgical intervention is not possible/safe
* Contraindication to MRI
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Hip Outcome Score | 8 months post randomisation (approximately 6 months post intervention)
  Hip Outcome Score is a patient reported outcome measure

SECONDARY OUTCOMES:
Patient Reported Outcome Measures | Regular intervals up to 38 months post randomisation (approximately 3 years post intervention)
Morphological and Physiological MRI | Regular intervals up to 38 months post randomisation (approximately 3 years post intervention)
  * Morphological Parameters
  * Measures of Osteoarthritis
Hip Radiographs | Regular intervals up to 38 months post randomisation (approximately 3 years post intervention)
  * Morphological Parameters
  * Measures of Osteoarthritis
Serum and Urinary Biomarkers of Osteoarthritis | Regular intervals up to 38 months post randomisation (approximately 3 years post intervention)
Clinical Examination | Regular intervals up to 38 months post randomisation (approximately 3 years post intervention)
  * Range of Movement
  * Impingement Tests

CONTACTS AND LOCATIONS:
Overall Officials: Sion Glyn-Jones, MA MBBS FRCS DPhil, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Nuffield Orthopaedic Centre, Oxford University Hospitals Trust, Oxford
  - Royal Berkshire Hospital, Reading

REFERENCES:
- [Derived] Palmer A, Fernquest S, Rombach I, Harin A, Mansour R, Dutton S, Dijkstra HP, Andrade T, Glyn-Jones S; FAIT Study Group. Medium-term results of arthroscopic hip surgery compared with physiotherapy and activity modification for the treatment of femoroacetabular impingement syndrome: a multi-centre randomised controlled trial. Br J Sports Med. 2025 Jan 2;59(2):109-117. doi: 10.1136/bjsports-2023-107712. PMID 39592214
- [Derived] Palmer AJR, Ayyar Gupta V, Fernquest S, Rombach I, Dutton SJ, Mansour R, Wood S, Khanduja V, Pollard TCB, McCaskie AW, Barker KL, Andrade TJMD, Carr AJ, Beard DJ, Glyn-Jones S; FAIT Study Group. Arthroscopic hip surgery compared with physiotherapy and activity modification for the treatment of symptomatic femoroacetabular impingement: multicentre randomised controlled trial. BMJ. 2019 Feb 7;364:l185. doi: 10.1136/bmj.l185. PMID 30733197
- [Derived] Palmer AJ, Ayyar-Gupta V, Dutton SJ, Rombach I, Cooper CD, Pollard TC, Hollinghurst D, Taylor A, Barker KL, McNally EG, Beard DJ, Andrade AJ, Carr AJ, Glyn-Jones S. Protocol for the Femoroacetabular Impingement Trial (FAIT): a multi-centre randomised controlled trial comparing surgical and non-surgical management of femoroacetabular impingement. Bone Joint Res. 2014 Nov;3(11):321-7. doi: 10.1302/2046-3758.311.2000336. PMID 25431439